CLINICAL TRIAL: NCT02514447
Title: Phase 1b/2a Safety and Pharmacokinetic Study of G1T28 in Patients With Previously Treated Extensive Stage Small Cell Lung Cancer (SCLC) Receiving Topotecan Chemotherapy
Brief Title: Trilaciclib (G1T28) in Patients With Previously Treated Extensive Stage SCLC Receiving Topotecan Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G1T28-03; 2016-004611-13 (EudraCT Number)
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Results first posted 2022-06-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; CDK4/6 Inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — trilaciclib; Topotecan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b (Experimental): Patients in Parts 2a and 2b were randomized 1:2 to placebo. Patients received placebo administered IV once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of placebo on Days 1 to 5, patients received IV topotecan (1.5 mg/m²).
  Interventions: Drug: Placebo; Drug: Topotecan
- Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a (Experimental): Patients in Part 2a were randomized 2:1 to trilaciclib. Patients received trilaciclib (240 mg/m²) administered IV once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b (Experimental): Patients in Part 2b were randomized 2:1 to trilaciclib. Patients received trilaciclib (240 mg/m²) administered IV once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (1.5 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 (Experimental): Patients received trilaciclib (200 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (1.50 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 (Experimental): Patients received trilaciclib (200 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (1.25 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 (Experimental): Patients received trilaciclib (200 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 (Experimental): Patients received trilaciclib (240 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 (Experimental): Patients received trilaciclib (280 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan
- Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1 (Experimental): Patients received trilaciclib (240 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (1.0 mg/m²).
  Interventions: Drug: Trilaciclib; Drug: Topotecan

INTERVENTIONS:
Drug: Trilaciclib
  Other Names: G1T28; CDK 4/6 inhibitor
  Arms: Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1; Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1; Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1; Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1; Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a; Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1; Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b; Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1
Drug: Placebo
  Arms: Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b
Drug: Topotecan

SUMMARY:
This was a study to investigate the potential clinical benefit of trilaciclib (G1T28), a Cyclin Dependent Kinase (CDK) 4/6 inhibitor, in preserving the bone marrow and the immune system, in order to decrease chemotherapy-induced myelosuppression and improve anti-tumor efficacy when administered prior to topotecan in patients previously treated for extensive-stage SCLC.

The study consisted of 2 parts: a limited open-label, dose-finding portion (Part 1), and a randomized double-blind portion (Part 2). Both parts included 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase began on the day of first dose with study treatment and completes at the Post-Treatment Visit.

DETAILED DESCRIPTION:
Overall, up to 130 patients were planned to be enrolled in the study. In Part 1, approximately 40 patients were planned to be enrolled, assuming 9 to 10 cohorts. Part 1 was open-label, and no randomization or blinding was required. In Part 2A, approximately 45 patients were to be enrolled and randomly assigned (2:1) to trilaciclib (240 mg/m2) and topotecan (0.75 mg/m2) or placebo and topotecan (1.5 mg/m2). In Part 2B, approximately 45 patients were to be enrolled and randomly assigned (2:1) to trilaciclib (240 mg/mg2) and topotecan (1.5 mg/m2) or placebo and topotecan (1.5 mg/m2).

Patients who received placebo in Part 2A and Part 2B were to be combined into a single placebo group for the analysis to compare with trilaciclib+topotecan 1.5 mg/m2 with placebo + topotecan 1.5 mg/m2 (proximately 30 per treatment group).

The sample size calculation was to demonstrate the superiority of trilaciclib + topotecan 1.5 mg/m2 over placebo + topotecan 1.5 mg/m2 with respect to at least 1 of the primary endpoints. The overall type I error rate was 1-sided 0.10. Using the most conservative Bonferroni procedure for the 2 primary endpoints, a 1-sided individual type I error rate 0.10/2=0.05 was assigned to each outcome variable (DSN in Cycle 1 and occurrence of SN) in the sample size calculation. Assuming a common standard deviation of 2.5, a difference in the duration of SN in Cycle 1 of at least 2 days between the treatment groups, a sample size of 28 per arm was required to have 90% power to detect the assumed treatment effect. For occurrence of SN, assuming the event rate was 45% for placebo group, to detect an absolute reduction of 37% by trilaciclib group with 90% power would require a sample size of at least 29 per arm. Thus, 30 per arm was needed to ensure 90% power to detect assumed treatment effect for DSN in Cycle 1 and occurrence of SN. All calculations were carried out using the POWER procedure in SAS®, Version 9.4 procedure in SAS®, Version 9.4 or higher.

The results from endpoints that were commonly collected at Part 1 and part 2 are presented together in this report.

The posted results represent the final results of Study G1T28-03, a Phase 1b/2a safety and pharmacokinetic (PK) study of trilaciclib (G1T28) in patients with previously treated extensive-stage small cell lung cancer (SCLC) receiving topotecan chemotherapy in the second/third-line (2/3L) setting. The final myelopreservation efficacy results for both parts and exposure for Part 1 are from database lock 1 (data cut-off [DCO] for Primary Completion Date [PCD] 28 September 2018). The final anti-tumor efficacy (BOR, DOR, PFS) for both parts, final overall survival for Part 1 and exposure data from Part 2 are from a second database lock 2 (DCO 31 May 2019) and the final overall survival for Part 2 and safety (adverse events) are through the end of the study on October 4, 2021 which resulted in the final database lock (DCO 01 Nov 2021).

The maximum time frames provided reflect the time from when the first patient could be evaluated for an endpoint (ie. date of first dose of first patient) to the time when the data from both parts presented for that endpoint was considered final.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects aged ≥18 years
* Confirmed diagnosis of SCLC by histology or cytology, preferably including the presence of neuroendocrine features by immunohistochemistry
* Progression during or after prior first- or second-line chemotherapy and eligible to receive topotecan therapy
* At least 1 target lesion that is measurable by RECIST, Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Adequate organ function

Key Exclusion Criteria:

* Presence of brain metastases requiring immediate treatment with radiation therapy or steroids.
* Uncontrolled ischemic heart disease or uncontrolled symptomatic congestive heart failure
* Known history of stroke or cerebrovascular accident within 6 months prior to enrollment
* Other uncontrolled serious chronic disease or conditions that in the investigator's opinion could affect compliance or follow-up in the protocol
* Concurrent radiotherapy to any site or radiotherapy within 2 weeks prior to enrollment or previous radiotherapy to the target lesion sites
* Receipt of any systemic chemotherapy regimen within 4 weeks prior to enrollment or a noncytotoxic investigational medication within 2 weeks prior to enrollment
* History of topotecan treatment for SCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (50):
- United States (35):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Compassionate Cancer Care Medical Group, Inc., Corona, California
  - Sutter Medical Group, Sacramento, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Memorial Hospital - University of Colorado Health, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Colorado Health, Oncology Clinical Research Northern Region, Fort Collins, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, Tavares, Florida
  - University Cancer and Blood Center, LLC, Athens, Georgia
  - Emory University, Atlanta, Georgia
  - Northside Hospital - Georgia Cancer Specialists, Atlanta, Georgia
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - North Shore Hematology Oncology Associates PC, East Setauket, New York
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Oklahoma University - Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Hanna Cancer Associates - University of Tennessee, Knoxville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - M.D. Anderson, Houston, Texas
  - Millennium Oncology, Houston, Texas
  - Southwest Cancer Center, Lubbock, Texas
  - Texas Oncology, Tyler, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- AZ Klina, Brasschaat, Belgium
- Bosnia and Herzegovina (2):
  - University Clinical Centre Banja Luka, Banja Luka
  - University Clinical Centre Sarajevo, Sarajevo
- Croatia (3):
  - Clinical Hospital Centre Osijek, Osijek
  - University Clinical Hospital Centre " Sestre Milosrdnice", Zagreb
  - University Hospital Centre Zagreb, Clinic For Pulmonary Diseases Jordanovac, Zagreb
- University Clinic of Radiotherapy and Oncology Skopje, Skopje, North Macedonia
- Serbia (5):
  - Clinic for Pulmology, Clinical Centre of Serbia, Belgrade
  - Clinical Hospital Centre Bezanijska Kosa, Belgrade
  - Oncology and Radiology Institute of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina Clinic for Thoracic Oncology, Kamenitz
  - Clinical Center Nis, Clinic for Lung Diseases, Niš
- Slovakia (2):
  - VOU Department of Radiotherapy and Oncology, Košice
  - POKO POPRAD, s.r.o., Poprad
- University Clinic of Respiratory and Allergic Diseases Golnik, Golnik, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hart LL, Ferrarotto R, Andric ZG, Beck JT, Subramanian J, Radosavljevic DZ, Zaric B, Hanna WT, Aljumaily R, Owonikoko TK, Verhoeven D, Xiao J, Morris SR, Antal JM, Hussein MA. Myelopreservation with Trilaciclib in Patients Receiving Topotecan for Small Cell Lung Cancer: Results from a Randomized, Double-Blind, Placebo-Controlled Phase II Study. Adv Ther. 2021 Jan;38(1):350-365. doi: 10.1007/s12325-020-01538-0. Epub 2020 Oct 29. PMID 33123968
- [Derived] Li C, Horton JK, Sale M, Curd L, Goti V, Tao W, Beelen A. Pharmacokinetic Drug-Drug Interaction Studies Between Trilaciclib and Midazolam, Metformin, Rifampin, Itraconazole, and Topotecan in Healthy Volunteers and Patients with Extensive-Stage Small-Cell Lung Cancer. Clin Drug Investig. 2022 Aug;42(8):679-692. doi: 10.1007/s40261-022-01179-x. Epub 2022 Jul 16. PMID 35842567
- [Derived] Hussein M, Maglakelidze M, Richards DA, Sabatini M, Gersten TA, Lerro K, Sinielnikov I, Spira A, Pritchett Y, Antal JM, Malik R, Beck JT. Myeloprotective Effects of Trilaciclib Among Patients with Small Cell Lung Cancer at Increased Risk of Chemotherapy-Induced Myelosuppression: Pooled Results from Three Phase 2, Randomized, Double-Blind, Placebo-Controlled Studies. Cancer Manag Res. 2021 Aug 9;13:6207-6218. doi: 10.2147/CMAR.S313045. eCollection 2021. PMID 34408488
- [Derived] Ferrarotto R, Anderson I, Medgyasszay B, Garcia-Campelo MR, Edenfield W, Feinstein TM, Johnson JM, Kalmadi S, Lammers PE, Sanchez-Hernandez A, Pritchett Y, Morris SR, Malik RK, Csoszi T. Trilaciclib prior to chemotherapy reduces the usage of supportive care interventions for chemotherapy-induced myelosuppression in patients with small cell lung cancer: Pooled analysis of three randomized phase 2 trials. Cancer Med. 2021 Sep;10(17):5748-5756. doi: 10.1002/cam4.4089. Epub 2021 Aug 18. PMID 34405547
- [Derived] Li C, Hart L, Owonikoko TK, Aljumaily R, Rocha Lima CM, Conkling PR, Webb RT, Jotte RM, Schuster S, Edenfield WJ, Smith DA, Sale M, Roberts PJ, Malik RK, Sorrentino JA. Trilaciclib dose selection: an integrated pharmacokinetic and pharmacodynamic analysis of preclinical data and Phase Ib/IIa studies in patients with extensive-stage small cell lung cancer. Cancer Chemother Pharmacol. 2021 May;87(5):689-700. doi: 10.1007/s00280-021-04239-9. Epub 2021 Feb 17. PMID 33595690
- See also: Myelopreservation with Trilaciclib in Patients Receiving Topotecan for Small Cell Lung Cancer: Results from a Randomized, Double-Blind, Placebo-Controlled Phase II Study — https://pubmed.ncbi.nlm.nih.gov/33123968/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b: Patients in Parts 2a and 2b were randomized 1:2 to placebo. Patients received placebo administered IV once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of placebo on Days 1 to 5, patients received IV topotecan (1.5 mg/m²).
  Placebo
  Topotecan
- Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a: Patients in Part 2a were randomized 2:1 to trilaciclib. Patients received trilaciclib (240 mg/m²) administered IV once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75 mg/m²).
  Trilaciclib
  Topotecan
- Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b: Patients in Part 2b were randomized 2:1 to trilaciclib. Patients received trilaciclib (240 mg/m²) administered IV once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (1.5 mg/m²).
  Trilaciclib
  Topotecan
Period: Overall Study
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Started | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 24 | 28 | 29 | 0 | 3 | 4 | 8 | 6 | 5
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Termination of Study | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study completion per Investigator | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b: Patients in Parts 2a and 2b were randomized 1:2 to placebo. Patients received placebo administered IV once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of placebo on Days 1 to 5, patients received IV topotecan (1.5 mg/m²).
  Placebos
  Topotecan
- Total: Total of all reporting groups
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1 | Total
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 20 | 1 | 1 | 1 | 6 | 4 | 2 | 71
  >=65 years | 11 | 12 | 12 | 1 | 2 | 3 | 2 | 3 | 6 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (8.1) | 63 (8.2) | 62 (7.3) | 66 (9.2) | 69 (9.1) | 71 (6.1) | 62 (8.4) | 63 (8.9) | 69 (10.4) | 64 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 10 | 0 | 2 | 0 | 5 | 0 | 4 | 52
  Male | 12 | 16 | 22 | 2 | 1 | 4 | 3 | 7 | 4 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 30 | 31 | 2 | 3 | 4 | 8 | 7 | 8 | 121
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 6
  White | 26 | 29 | 30 | 2 | 3 | 4 | 7 | 6 | 7 | 114
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 27 | 14 | 2 | 3 | 4 | 8 | 7 | 8 | 91
  Serbia | 11 | 3 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 26
  Belgium | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  North Macedonia | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Croatia | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  Grade 0= Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Grade 2= Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    Grade 0-1 | 27 | 27 | 29 | 2 | 3 | 4 | 6 | 7 | 7 | 112
    Grade 2 | 2 | 3 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 11
Body Weight at Screening [Mean (Standard Deviation); unit: kg] | 72.7 (16.37) | 71.9 (17.08) | 75.7 (17.28) | 95.2 (22.20) | 72.6 (23.59) | 90.1 (23.05) | 73.5 (29.88) | 86.3 (19.25) | 67.8 (15.00) | 74.7 (18.55)
Height at Screening [Mean (Standard Deviation); unit: cm] | 166.2 (9.85) | 169.0 (9.49) | 172.2 (10.01) | 176.2 (1.27) | 169.7 (18.53) | 175.3 (5.42) | 165.2 (12.93) | 175.3 (3.49) | 167.4 (16.74) | 169.5 (10.56)
BMI at Screening [Mean (Standard Deviation); unit: kg/m^2] | 26.13 (4.239) | 25.04 (4.820) | 25.43 (5.113) | 30.72 (7.595) | 24.63 (2.430) | 29.05 (6.218) | 26.06 (7.164) | 28.11 (6.232) | 24.15 (3.502) | 25.79 (4.984)
Body Surface Area at Screening [Mean (Standard Deviation); unit: m^2] | 1.80 (0.234) | 1.81 (0.234) | 1.88 (0.234) | 2.11 (0.200) | 1.83 (0.398) | 2.05 (0.282) | 1.79 (0.398) | 2.01 (0.185) | 1.76 (0.274) | 1.85 (0.255)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe (Grade 4) Neutropenia in Cycle 1
Description: Duration of severe neutropenia (DSN; days) was defined as the number of days from the date of the first ANC value of <0.5 × 10^9/L observed between start of cycle and end of cycle to the date of the first ANC value ≥0.5 × 10^9/L that met the following criteria: (1) occurred after the ANC value of <0.5 × 10^9/L and (2) no other ANC values <0.5 × 10^9/L occurred between this day and end of cycle. DSN is set to 0 for patients who did not experience SN in a cycle, including those who were randomized but never treated. Data from unscheduled visits and the actual assessment date (rather than visit date) were included in the derivation.
Time Frame: Evaluated for Cycle 1 (i.e., from date of first dose of study drug (Part 1)/randomization (Part 2) to the end of Cycle 1, each cycle = 21 days)
Population: The intent-to-treat (ITT) analysis set: All enrolled patients who received at least one dose of study drugs in Part 1 and all randomized patients in Part 2 on the basis of the assigned treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
days | 8 (6.0) | 1 (3.1) | 2 (3.9) | 14 (1.4) | 8 (6.8) | 0 (0) | 0 (0) | 2 (3.6) | 3 (5.5)
Statistical Analysis 1: Comparison: Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b vs Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b; Analysis was for Part 2 data: Treatment difference was evaluated using a nonparametric analysis of covariance (ANCOVA). The nonparametric ANCOVA included study baseline ANC value as covariate, stratification factors of ECOG performance status (0 to 1 versus 2) and sensitivity to first line treatment (sensitive or resistant) and treatment as fixed effects; Test type: Superiority; p < 0.0001, non-parametric ANCOVA — A Hochberg-based gatekeeping procedure was used to control the global familywise error rate across the multiple null hypotheses (primary and key secondary myelosuppression efficacy endpoints) in a strong sense at a 1-sided 0.10 level; Hochberg-based gatekeeping procedure

2. Primary Outcome: Occurrence of Severe (Grade 4) Neutropenia
Description: Number of Participants with severe (Grade 4) neutropenia (SN) was a binary variable. If a patient had at least 1 absolute neutrophil count value <0.5 × 10^9/L during the Treatment Period, the patient was assigned as Yes to the occurrence of SN; otherwise, it was No.
Time Frame: During the treatment period. From date of first dose (Part 1)/randomization (Part 2), 21 day treatment cycles continue until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator (assessed up to 1090 days).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 22 | 5 | 13 | 2 | 2 | 1 | 0 | 2 | 3
Statistical Analysis 1: Comparison: Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b vs Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b; The occurrence of SN was a binary variable. Treatment group difference was analyzed using modified Poisson regression to account for the variable duration of the Treatment Period for each patient. The model included baseline ANC as a covariate, stratification factors of ECOG performance status (0 or 1 vs 2), sensitivity to 1st line treatment (sensitive or resistant), and treatment as fixed effects. The logarithm transformation of # of cycles was included as an offset variable in the modeling; Test type: Superiority; p = 0.0160, Modified Poisson — [p-value comment as in outcome 1, analysis 1]; Hochberg-based gatekeeping procedure

3. Primary Outcome: Assess the Dose Limiting Toxicities (DLTs) of G1T28/Trilaciclib Administered With Topotecan in Part 1
Description: The percentage of patients experiencing DLTs in Part 1 of the study in each cohort, including:
  * Absolute neutrophil count (ANC) < 0.5 × 10^9/L lasting for ≥ 7 days
  * ≥ Grade 3 neutropenic infection/febrile neutropenia
  * Grade 4 thrombocytopenia or ≥ Grade 3 thrombocytopenia with bleeding
  * Unable to start next cycle of chemotherapy due to lack of recovery to an ANC ≥ 1.5 × 10^9/L and platelet count ≥ 100 × 10^9/L; a delay of up to 1 week from the scheduled start of Cycle 2 is allowed for recovery of ANC and platelet count, and is not considered a DLT
  * ≥ Grade 3 nonhematologic toxicity (nausea, vomiting, and diarrhea failing maximal medical management; fatigue lasting for > 72 hours)
Time Frame: Evaluated for Cycle 1 (i.e., from date of first dose of study drug (Part 1) to the end of Cycle 1, each cycle = 21 days)
Population: The safety analysis set: All enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m²- Part 1 Cohort 1; Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m²- Part 1 Cohort 2; Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m²- Part 1 Cohort 3; Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m²- Part 1 Cohorts 4 and 6; Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m²- Part 1 Cohort 5; Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m²- Part 1 Cohort 7: Patients received trilaciclib (200, 240, or 280 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75, 1.0, 1.25, or 1.50 mg/m²).
  Trilaciclib
  Topotecan
Arm/Group | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m²- Part 1 Cohort 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m²- Part 1 Cohort 2 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m²- Part 1 Cohort 3 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m²- Part 1 Cohorts 4 and 6 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m²- Part 1 Cohort 5 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m²- Part 1 Cohort 7
Number analyzed (Participants) | 2 | 3 | 4 | 8 | 7 | 8
Participants | 2 | 2 | 2 | 0 | 2 | 2

4. Secondary Outcome: Pharmacokinetic Profile for Trilaciclib (G1T28) When Administered With Topotecan
Description: Maximum concentration (Cmax) of trilaciclib (G1T28) when administered with topotecan
Time Frame: Part 1 of the study during Cycle 1 Day 4 : predose, 0.5, 1, 1.5, 2, 2.5, 3, 4.5, 6.5, 8.5 (optional), and 24.5 hours post dose. Part 2 of the study during Cycle 1 Day 4 : predose, 0.5, 1, between 3 to 4 hours and between 5.5 to 6.5 hours post dose.
Population: All patients who had evaluable PK profiles for both treatments and analytes.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Trilaciclib (G1T28) 200 mg/m² + Topotecan - Part 1; Trilaciclib (G1T28) 240 mg/m² + Topotecan - Part 1; Trilaciclib (G1T28) 280 mg/m² + Topotecan - Part 1: Patients received trilaciclib (200, 240, or 280 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75, 1.0, 1.25, or 1.50 mg/m²).
  Trilaciclib
  Topotecan
Arm/Group | Trilaciclib (G1T28) 200 mg/m² + Topotecan - Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan - Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan - Part 1 | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b
Number analyzed (Participants) | 9 | 15 | 7 | 0 | 28 | 30
ng/ml | 1060 (59.0) | 1220 (120) | 2220 (75.2) |  | 913 (59.6) | 1100 (54.8)

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Median time (months) and 95% CI from date of first dose of study drug/randomization until date of documented disease progression or death due to any cause.
  Investigators followed the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 guidelines for tumor assessments to determine progression. Progressive Disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From date of first dose of study drug (Part 1)/randomization (Part 2), until date of documented disease progression or death due to any cause (evaluated up to a maximum of 1335 days).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
months | 4.2 [1.6 to 6.2] | 3.0 [1.7 to 3.6] | 4.2 [2.1 to 5.2] | 5.5 [NA to NA] — Due to only 1 event, the confidence limits for the median could not be estimated. | 4.3 [1.4 to 8.9] | 3.6 [2.1 to 4.2] | 4.5 [0.7 to 5.9] | 1.8 [1.3 to 6.9] | 2.1 [1.4 to 7.5]

6. Secondary Outcome: Overall Survival (OS)
Description: Median time (months) and 95% CI from date of first dose date of study drug/randomization until date of death. Patients who do not die during the study will be censored at the date last known to be alive.
Time Frame: From date of first dose of study drug (Part 1)/randomization (Part 2) until the date of death due to any cause (evaluated up to a maximum of 2220 days).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
months | 6.5 [3.5 to 11.3] | 5.8 [4.1 to 8.1] | 6.2 [4.0 to 9.9] | NA [NA to NA] — Due to zero events, the median and its confidence limits could not be estimated. | 10.6 [8.3 to 25.3] | 8.3 [4.5 to 11.8] | 9.4 [1.1 to 12.5] | 4.4 [2.1 to 10.0] | 10.0 [2.1 to NA] — The upper confidence limit for the median was not estimable, as the upper confidence limits for the survivor function lies above 0.5.

7. Secondary Outcome: Assess the Hematologic Profile of G1T28/Trilaciclib Administered With Topotecan
Description: The weekly event rate of Major Adverse Hematologic Events (MAHE) events
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: events per participant/week
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
events per participant/week | 0.258 | 0.091 | 0.102 | 0.403 | 0.156 | 0.102 | 0.037 | 0.085 | 0.073

8. Secondary Outcome: Tumor Response Based on RECIST, Version 1.1
Description: The percentage of patients who fall into each category of Best overall response (BOR) as defined by RECIST, Version 1.1.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  When no imaging/measurement is done, the patient is not evaluable (NE); and if only a subset of lesion measurements are made, usually the case is also considered NE.
Time Frame: From date of first dose of study drug (Part 1)/randomization (Part 2) until the occurrence of progressive disease, withdrawal of consent, or initiation of subsequent anti-cancer therapy, (assessed up to a maximum of 1335 days).
Population: Response-Evaluable analysis set: All patients who are in the mITT, have measurable disease (target lesions) at the baseline tumor assessment, and either (i) have at least 1 post-baseline tumor assessment, (ii) have clinical progression as noted by the investigator before their first post-baseline tumor scan, or (iii) have died due to disease progression before their first post-baseline tumor scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 26 | 29 | 30 | 2 | 3 | 4 | 8 | 6 | 7
Participants
  Complete Response (CR) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 5 | 3 | 5 | 1 | 2 | 0 | 1 | 0 | 1
  Stable Disease (SD) | 10 | 15 | 13 | 1 | 0 | 3 | 6 | 3 | 3
  Progressive Disease (PD) | 6 | 9 | 6 | 0 | 1 | 1 | 1 | 2 | 2
  Not Evaluable (NE) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No post-baseline tumor assessment (Missing) | 2 | 2 | 6 | 0 | 0 | 0 | 0 | 1 | 1

9. Secondary Outcome: Occurrence of RBC Transfusions
Description: Percentage of patients requiring a RBC transfusion on/after week 5
Time Frame: During the treatment period. From date of first dose (Part 1)/randomization (Part 2), 21 day treatment cycles continue until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator (assessed up to 1056 days).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 12 | 5 | 10 | 2 | 1 | 2 | 1 | 1 | 2

10. Secondary Outcome: Need for Treatment With Hematopoietic Growth Factors
Description: Percentage of patients requiring G-CSF administration.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 19 | 8 | 16 | 2 | 2 | 1 | 4 | 2 | 3

11. Secondary Outcome: Chemotherapy Cycles and Modifications Overall
Description: Average exposure and cycle modifications in chemotherapy (topotecan)
Time Frame: During the treatment period. From date of first dose, 21 day treatment cycles continue until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator (assessed up to a maximum of 1335 days).
Population: Safety analysis set: All enrolled patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 28 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
cycles
  Number of cycles completed | 4 (3.4) | 5 (5.4) | 5 (4.4) | 6 (0.0) | 7 (5.0) | 4 (1.7) | 6 (2.9) | 4 (3.4) | 4 (2.2)
  Number of cycles delayed | 1 (1.2) | 2 (2.5) | 1 (1.4) | 3 (1.4) | 1 (1.2) | 1 (0.5) | 1 (0.8) | 0 (0.5) | 1 (1.0)

12. Secondary Outcome: Pharmacokinetic Profile for Topotecan When Administered With Trilaciclib (G1T28)
Description: Maximum concentration (Cmax) of topotecan when administered with trilaciclib (G1T28)
Time Frame: as for outcome 4
Population: All patients who had evaluable PK profiles for both treatments and analytes.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Trilaciclib (G1T28) + Topotecan 0.75 mg/m²- Part 1; Trilaciclib (G1T28) + Topotecan 1 mg/m²- Part 1; Trilaciclib (G1T28) + Topotecan 1.25 mg/m²- Part 1: Patients received trilaciclib (200, 240, or 280 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (0.75, 1.0, 1.25, or 1.50 mg/m²).
  Trilaciclib
  Topotecan
- Trilaciclib (G1T28) + Topotecan 1.50 mg/m²- Part 1: Patients received trilaciclib (200, 240, or 280 mg/m²) administered intravenously (IV) once daily on Days 1 to 5 of each 21-day topotecan chemotherapy cycle.
  Following administration of trilaciclib on Days 1 to 5, patients received IV topotecan (1.50 mg/m²).
Arm/Group | Trilaciclib (G1T28) + Topotecan 0.75 mg/m²- Part 1 | Trilaciclib (G1T28) + Topotecan 1 mg/m²- Part 1 | Trilaciclib (G1T28) + Topotecan 1.25 mg/m²- Part 1 | Trilaciclib (G1T28) + Topotecan 1.50 mg/m²- Part 1 | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b
Number analyzed (Participants) | 19 | 7 | 3 | 2 | 25 | 27 | 29
ng/ml | 21.1 (34.6) | 36.8 (41.8) | 52.4 (66.5) | NA (NA) — There was an insufficient number of participants with evaluable PK profiles to calculate the Cmax geometric mean or median for the Part 1 Topotecan 1.5 mg/m2 cohort. | 43.0 (39.0) | 17.5 (36.5) | 41.4 (46.9)

13. Secondary Outcome: Duration of Response (DOR)
Description: The median months and 95% CIs of duration of response.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 6 | 3 | 5 | 1 | 2 | 0 | 1 | 0 | 1
months | 4.9 [2.1 to NA] — The upper confidence limit for the median was not estimable, due to an insufficient number of participants with events, as the upper confidence limits for the survivor function lies above 0.5. | 7.8 [4.1 to NA] — The upper confidence limit for the median was not estimable, due to an insufficient number of participants with events, as the upper confidence limits for the survivor function lies above 0.5. | 6.8 [2.8 to NA] — The upper confidence limit for the median was not estimable, due to an insufficient number of participants with events, as the upper confidence limits for the survivor function lies above 0.5. | NA [NA to NA] — Due to an insufficient number of participants with events, zero or only 1 event, the confidence limits for the median could not be estimated. | 5.4 [3.1 to 7.7] |  | 6.7 [NA to NA] — The upper confidence limit for the median was not estimable, due to an insufficient number of participants with events, as the upper confidence limits for the survivor function lies above 0.5. |  | NA [NA to NA] — Due to an insufficient number of participants with events, zero or only 1 event, the confidence limits for the median could not be estimated.

14. Secondary Outcome: Occurrence of Intravenous (IV) Antibiotic Use
Description: Percentage of patients requiring systemic/IV antibiotics
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 8 | 8 | 7 | 2 | 1 | 1 | 1 | 2 | 1

15. Secondary Outcome: Occurrence of Platelet Transfusions
Description: Percentage of patients requiring a platelet transfusion
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 9 | 4 | 8 | 0 | 1 | 0 | 0 | 1 | 0

16. Secondary Outcome: Occurrence of Febrile Neutropenia Adverse Events
Description: Percentage of patients who experience febrile neutropenia adverse events
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 5 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0

17. Secondary Outcome: Occurrence of Infection Serious Adverse Events (SAEs)
Description: Percentage of patients experiencing an SAE that codes to the Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) of Infections and Infestations
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 3 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 1

18. Secondary Outcome: Occurrence of Pulmonary Infection Serious Adverse Events (SAEs)
Description: Percentage of patients experiencing an SAE that codes to the Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) of Infections and Infestations and falls into a preferred term (PT) categorized as a pulmonary infection custom MedDRA query (CMQ)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1

19. Secondary Outcome: Dose Reductions in Chemotherapy (Topotecan)
Description: Overall event rate of dose reductions in chemotherapy (topotecan)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: events per participant per cycle
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
events per participant per cycle | 0.116 | 0.053 | 0.051 | 0.500 | 0.250 | 0.118 | 0.089 | 0.040 | 0.036

20. Secondary Outcome: Occurrence of Grade 3 and 4 Hematologic Toxicities
Description: The count of patients with any hematologic lab value that meets the CTCAE toxicity grade criteria for ≥ Grade 3 and the value is treatment emergent (occurs after first dose of study drug). Labs include: Hemoglobin (HGB), hematocrit, white blood cell (WBC), platelet counts, ANC, ALC, Monocyte Absolute, Basophil Absolute, and Eosinophil Absolute.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 27 | 25 | 29 | 2 | 3 | 4 | 7 | 7 | 7

21. Secondary Outcome: Occurrence of Grade 4 and Grade 3/4 Decreased Platelet Count Laboratory Values (Thrombocytopenia)
Description: The count of patients with any platelet lab value that meets the CTCAE toxicity grade criteria for ≥ Grade 3 and the value is treatment emergent (occurs after first dose of study drug).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants
  Overall Grade 3/4 Thrombocytopenia | 19 | 15 | 21 | 2 | 2 | 3 | 2 | 4 | 4
  Overall Grade 4 Thrombocytopenia | 11 | 9 | 13 | 2 | 1 | 2 | 0 | 2 | 1

22. Secondary Outcome: Occurrence of Erythropoietin-stimulating Agent (ESA) Administrations
Description: The count of patients who received any ESA administration.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 29 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
Participants | 6 | 5 | 1 | 2 | 1 | 0 | 1 | 0 | 1

23. Secondary Outcome: Chemotherapy Exposure
Description: Average duration of exposure to chemotherapy (topotecan) in days.
Time Frame: as for outcome 11
Population: Safety analysis set: All enrolled patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
Number analyzed (Participants) | 28 | 30 | 32 | 2 | 3 | 4 | 8 | 7 | 8
days | 94 (75.9) | 110 (132.1) | 109 (97) | 147 (9.9) | 147 (116.9) | 102 (38.9) | 124 (65.8) | 78 (74.9) | 83 (51.8)

ADVERSE EVENTS:
Time Frame: The SAE reporting period started at the time of informed consent and the AE reporting period started from the time of first dose of study drug; both were assessed through 30 calendar days after the last administration of trilaciclib (G1T28) + topotecan (assessed up to a maximum of 1689 days). All-Cause Mortality was assessed from the date of first dose of study drug (Part 1)/randomization (Part 2) until the date of death due to any cause (evaluated up to a maximum of 2196 days).
Description: The safety analysis set (AEs and SAEs) includes all enrolled patients who received at least 1 dose of study drug (topotecan or trilaciclib/placebo). Analyses using the safety analysis set will be conducted on the basis of the actual treatment received.
  The intent-to-treat (ITT) analysis set (All-Cause Mortality) includes all enrolled patients who received at least one dose of study drugs in Part 1 and all randomized patients in Part 2 on the basis of the assigned treatment.
Arm/Group | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1
All-Cause Mortality (participants affected / at risk) | 24/29 | 28/30 | 29/32 | 0/2 | 3/3 | 4/4 | 8/8 | 6/7 | 5/8
Serious Adverse Events (participants affected / at risk) | 7/28 | 15/30 | 12/32 | 2/2 | 1/3 | 2/4 | 0/8 | 1/7 | 1/8
Other Adverse Events (participants affected / at risk) | 27/28 | 29/30 | 32/32 | 2/2 | 3/3 | 4/4 | 8/8 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b (N=28) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a (N=30) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b (N=32) | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 (N=2) | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 (N=3) | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 (N=4) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 (N=8) | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 (N=7) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1 (N=8)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 1 | 1 | 1 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary emobolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2 (2) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (2) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 (4) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 (7) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 (3) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Topotecan 1.5 mg/m² - Parts 2a and 2b (N=28) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Part 2a (N=30) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.5 mg/m² - Part 2b (N=32) | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.5 mg/m² - Cohort 1- Part 1 (N=2) | Trilaciclib (G1T28) 200 mg/m² + Topotecan 1.25 mg/m² - Cohort 2- Part 1 (N=3) | Trilaciclib (G1T28) 200 mg/m² + Topotecan 0.75 mg/m² - Cohort 3- Part 1 (N=4) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 0.75 mg/m² - Cohorts 4 and 6- Part 1 (N=8) | Trilaciclib (G1T28) 280 mg/m² + Topotecan 0.75 mg/m² - Cohort 5- Part 1 (N=7) | Trilaciclib (G1T28) 240 mg/m² + Topotecan 1.0 mg/m² - Cohort 7- Part 1 (N=8)
Neutropenia (Blood and lymphatic system disorders) | 23 (101) | 18 (58) | 24 (96) | 2 (19) | 3 (32) | 2 (7) | 5 (7) | 5 (14) | 5 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (96) | 17 (65) | 20 (133) | 2 (47) | 3 (37) | 3 (18) | 1 (4) | 4 (17) | 3 (26)
Anaemia (Blood and lymphatic system disorders) | 24 (94) | 14 (55) | 17 (57) | 2 (35) | 3 (36) | 2 (5) | 3 (39) | 4 (11) | 6 (24)
Leukopenia (Blood and lymphatic system disorders) | 9 (36) | 7 (14) | 4 (7) | 2 (38) | 3 (54) | 1 (12) | 2 (35) | 2 (16) | 3 (49)
Fatigue (General disorders) | 10 (16) | 16 (22) | 13 (15) | 2 (3) | 3 (4) | 2 (2) | 4 (5) | 1 (3) | 4 (8)
Pyrexia (General disorders) | 5 (6) | 2 (2) | 8 (8) | 1 (2) | 0 | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (4) | 5 (8) | 2 (3) | 2 (2) | 1 (1) | 1 (2) | 0 | 2 (6) | 2 (3)
Non-cardiac chest pain (General disorders) | 0 | 7 (9) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 2 (3)
Oedema peripheral (General disorders) | 0 | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0
Chest pain (General disorders) | 0 | 3 (3) | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0
Chills (General disorders) | 2 (3) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 (21) | 16 (20) | 9 (18) | 0 | 3 (3) | 2 (3) | 3 (3) | 4 (7) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (13) | 7 (7) | 5 (7) | 1 (1) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (5)
Vomiting (Gastrointestinal disorders) | 9 (11) | 4 (7) | 2 (7) | 0 | 1 (1) | 1 (1) | 2 (3) | 0 | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 4 (4) | 2 (2) | 2 (2) | 2 (2) | 0 | 2 (2) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (8) | 1 (2) | 0 | 1 (2) | 1 (1) | 1 (1) | 0 | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 (7) | 6 (7) | 6 (7) | 0 | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 6 (15) | 3 (8) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 3 (3) | 7 (8) | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (6) | 4 (7) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (4) | 0 | 0 | 0 | 1 (4) | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 (2) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 8 (10) | 3 (3) | 2 (3) | 1 (3) | 1 (1) | 5 (8) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (7) | 3 (3) | 0 | 1 (1) | 1 (1) | 4 (5) | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (4) | 0 | 1 (1) | 0 | 1 (1) | 2 (3) | 0 | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 | 1 (1) | 1 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 2 (3) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 | 0 | 0 | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (2) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 0 | 0 | 1 (3) | 0 | 0 | 0 | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 | 0 | 1 (1) | 0 | 2 (3) | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 (3) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 7 (9) | 4 (4) | 0 | 0 | 1 (1) | 3 (16) | 2 (13) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 4 (6) | 2 (2) | 2 (2) | 0 | 1 (1) | 3 (4) | 1 (3) | 2 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 | 1 (1) | 1 (1) | 0 | 0 | 1 (2)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 1 (3) | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 (6) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 (2) | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 | 0 | 1 (1) | 1 (2) | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 2 (2) | 0 | 0 | 1 (6) | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 3 (3) | 1 (1) | 0 | 0 | 1 (1) | 2 (13) | 1 (8) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 2 (3) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 | 1 (1) | 1 (1) | 0 | 0 | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 (2) | 2 (3) | 0 | 0 | 0 | 0 | 2 (2) | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Skin and subcutaneous tissue disorders) | 0 | 3 (3) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3 (3) | 0 | 1 (1) | 1 (2) | 0 | 1 (1) | 0 | 0
Hypotension (Vascular disorders) | 2 (3) | 5 (5) | 2 (3) | 1 (2) | 1 (1) | 0 | 0 | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 | 0 | 2 (3) | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 4 (4) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 (2) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0
Infusion site pain (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Infusion site reaction (General disorders) | 0 | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 0 | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 1 (2) | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (3) | 2 (2) | 2 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 2 (2) | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0
Dysphonia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 (2) | 0 | 1 (1) | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 1 (1) | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Face oedema (General disorders) | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 1 (1) | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Infusion site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Infusion site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Infusion site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (2) | 0
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 1 (4) | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0
Poor dental condition (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Blood immunoglobulin G decreased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Oral candidiasis (Infections and infestations) | 1 (1) | 0 | 1 (2) | 0 | 0 | 0 | 1 (1) | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 (4) | 0 | 0 | 0 | 0 | 1 (1) | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 1 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 (3) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Diplopia (Eye disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Eye discharge (Eye disorders) | 1 (1) | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
Limitation of the trial is small numbers of subjects, since it is a Phase 2 clinical trial.

Small sample size may have reduced the ability to observe statistically significant treatment effects on secondary myelopreservation measures (i.e. occurrence of FN AEs, infections and antibiotics usage).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT02514447/Prot_000.pdf
  • Statistical Analysis Plan: Region 1 (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT02514447/SAP_001.pdf
  • Statistical Analysis Plan: Region 2 (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT02514447/SAP_002.pdf